CLINICAL TRIAL: NCT01441804
Title: A Randomized Trial of 24-Week Versus 48-Week Courses of Peginterferon Plus Ribavirin for Patients With Genotype 1 Hepatitis C and IL28B CC Polymorphism
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Cai Qingxian, Third Affiliated Hospital, Sun Yat-Sen University, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAHG1IL-28BCC
Record Dates: First submitted 2011-09-24; First posted 2011-09-28 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 24-Week treatment group (Experimental): Genotype 1 chronic hepatitis C patients with IL28B CC Polymorphism and rapid virological response(undetectable HCV RNA at weeks 4) in this group will be treated with Peginterferon alfa-2a plus ribavirin for an additional 20 weeks
  Interventions: Drug: Peginterferon alfa2a; Drug: Ribavirin
- 48-Week treatment group (Active Comparator): Genotype 1 chronic hepatitis C patients with IL28B CC Polymorphism and rapid virological response(undetectable HCV RNA at weeks 4) in this group will be treated with Peginterferon alfa-2a plus ribavirin for an additional 44 weeks
  Interventions: Drug: Peginterferon alfa2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Peginterferon alfa2a — patients receive a dose of 180 µg of PEGASYS once a week for 24 weeks
  Arms: 24-Week treatment group
Drug: Ribavirin — patients receive a dose 800 to 1200 mg of ribavirin once a day(according to weight) for 24 weeks
  Arms: 24-Week treatment group
Drug: Peginterferon alfa2a — patients receive a dose of 180 µg of PEGASYS once a week for 48 weeks
  Arms: 48-Week treatment group
Drug: Ribavirin — patients receive a dose 800 to 1200 mg of ribavirin once a day(according to weight) for 48 weeks
  Arms: 48-Week treatment group

SUMMARY:
Patients with HCV genotype 1 and IL28B CC Polymorphism who have a rapid virological response to treatment are randomised to either 24 or 48 weeks HCV treatment. Our hypothesis is that there is no important difference in effect between the two treatment effect.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Serum Hepatitis C RNA > 10,000IU/mL
* Hepatitis C virus genotype 1
* IL28B CC polymorphism

Exclusion Criteria:

* Previous treatment for chronic Hepatitis C
* clinical or biological evidence of acute hepatitis, including serum ALT or AST > 300U/ml
* HIV antibody positive, hepatitis b surface antigen positive or known diagnosis of other chronic liver disease
* Contraindications to PR-based treatment:

  * Uncontrolled psychiatric illness
  * Active substance dependency
  * Known autoimmune disorder
  * Untreated thyroid disease
  * Uncontrolled seizure disorder
  * Pregnancy, lactation or inability to maintain contraception
  * Chronic kidney disease w/ estimated GFR< 60
  * ANC<1.5/nl, Hb<12g/dl, or platelets<75/nl
* Clinical or biochemical evidence of decompensated liver disease including:

  * History of encephalopathy
  * Ascites
  * Variceal bleeding
  * Bilirubin > 3g/dl or INR > 1.5
  * Life threatening disorder with expected median survival less than 5 years
  * Inability to comply with drug regimens or testing schedule required for study

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-05; Primary Completion 2014-05 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Sustained virological response (SVR) | 24 weeks after the end of treatment
  Undetectable HCVRNA in serum(<15IU/ml) 24 weeks after the end of treatment

SECONDARY OUTCOMES:
Change in health related quality as measured by short from 36 (SF-36) from baseline to 24 weeks after the end of treatment | baseline, 24 weeks after the end of treatment
Sick leave in patients treated for 24 or 48 weeks treatment | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gao Zhiliang, Doctor, Study Chair — The Third Affliated Hospital of Sun Yat-sen University; Zhao Zhixin, Doctor, Study Director — The Third Affliated Hospital of Sun Yat-sen University; Zhang Xiaohong, Doctor, Principal Investigator — The Third Affliated Hospital of Sun Yat-sen University
Locations (4):
- China (4):
  - The Eighth People's Hospital of Guangzhou, Guangzhou, Guangdong
  - The Third Affliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Panyu People's Hospital, Guangzhou, Guangdong
  - Zhongshan second people's hospital, Zhongshan, Guangdong